CLINICAL TRIAL: NCT03372902
Title: MSK Discovery Study: Use of cfNA To Distinguish Between Benign and Malignant BI-RADS 4 Radiographic Lesions
Brief Title: Development Of A Blood Test To Improve The Performance Of Breast Cancer Screening
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: GRAIL, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-598
Record Dates: First submitted 2017-12-11; First posted 2017-12-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Breast Benign
Keywords: Breast imaging; 17-598
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal mammograms (BI-RADS 1 or 2)
  Interventions: Device: Breast MRI; Device: Breast Mammogram; Other: Blood draw; Behavioral: online participant reported questionnaire
- suspicious lesion group (BI-RADS 4)
  Interventions: Device: Breast MRI; Device: Breast Mammogram; Other: Blood draw; Procedure: Breast Biopsy; Behavioral: online participant reported questionnaire

INTERVENTIONS:
Device: Breast MRI — Participants with dense breast tissue will get a mammogram and MRI
Device: Breast Mammogram — State-of-the-art full-field digital mammography (FFDM) and or digital breast tomosynthesis (DBT) comprising both raw and post-processed images as well as ultrasound and MRI images from the initial screening study will be collected and sent to the MSKCC Breast Radiology Department.
Other: Blood draw — Participants will donate approximately 60ml of peripheral blood. Mononuclear cells from peripheral blood will be used to extract germline DNA. Germline genomic testing will be employed as a matched control for tumor sequencing and for germline breast cancer susceptibility testing.
Procedure: Breast Biopsy — Tissue specimens from the biopsy of the BI-RADS 4 mammographic lesion and (among women undergoing surgical excision) the surgical specimen(s) will be subjected to genomic profiling at GRAIL, Inc. or MSKCC. The tumor specimens from the participants diagnosed with cancer during the follow-up period will also undergo molecular profiling.
  Groups: suspicious lesion group (BI-RADS 4)
Behavioral: online participant reported questionnaire — Participants will be asked to complete a questionnaire that covers the topics of breast health, general health and lifestyle, genetic testing, personal, and family history of cancer.

SUMMARY:
The purpose of this study is to collect blood and tissue to help develop tests that might be able to detect cancer earlier. The investigator will be collecting these samples and reviewing test results from participants who have had an area of concern found on breast imaging, as well as from participants who are scheduled to have a routine breast cancer screening mammogram.

ELIGIBILITY:
Inclusion Criteria:

* Females with one or more BI-RADS 4 radiographic lesions who are undergoing ultrasound, stereotactic or MRI-guided breast biopsy at MSKCC or at an MSK Alliance Member Site. If multiple imaging modalities were employed (mammogram, ultrasound, MRI) and no integrated score is provided, then the highest BI-RADS score will be used.
* Age ≥ 18 years at the time of breast biopsy
* Willing to provide blood samples for research purposes before biopsy.
* Able to provide written informed consent

Exclusion Criteria:

* Women with a BI-RADS 4 lesion who had the lesion previously biopsied
* Females with a current active malignancy other than non-melanoma skin cancers. Females are considered not to have a "current active" malignancy if they have completed therapy and have no evidence of systemic disease for at least three years from the initial diagnosis
* Currently pregnant women
* History of bilateral mastectomy.
* Participant has or is currently participating in another GRAIL-sponsored protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer
Study Population: Females with one or more BI-RADS 4 radiographic lesion who are undergoing ultrasound, stereotactic or MRI-guided breast biopsy at a participating study center.
Sampling Method: Non-Probability Sample
Enrollment: 628 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
number of participants with malignant biopsy | 2 years
  result of the biopsy of the BIRADS 4 breast

CONTACTS AND LOCATIONS:
Overall Officials: Katja Pinker-Domenig, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Hartford Healthcare Cancer Institute @ Hartford Hospital, Hartford, Connecticut
  - Baptist Alliance MCI, Miami, Florida
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm